CLINICAL TRIAL: NCT00473512
Title: A Phase I/II Open Label Study of the 17α-Hydroxylase/ C17,20 Lyase Inhibitor, Abiraterone Acetate in Patients With Prostate Cancer Who Have Failed Hormone Therapy
Brief Title: A Safety and Efficacy Study of Abiraterone Acetate in Participants With Prostate Cancer Who Have Failed Hormone Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016909; COU-AA-001 (Other: Cougar Biotechnology)
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Results first posted 2013-08-29 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Prostatic Neoplasms
Keywords: Abiraterone acetate; CB7630; Prostatic neoplasms; Hormone refractory prostate cancer; Castration resistant prostate cancer; Castration refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abiraterone acetate (Experimental): Abiraterone acetate 250 mg up to a maximum of 2000 mg capsules will be given orally daily for 28-day treatment period to determine the MTD in Phase 1 of the study. Participants will receive MTD of abiraterone acetate for 12 cycles (28 day each) in Phase 2 of the study. Dexamethasone 0.5 mg will be given orally (If participants have disease progression) daily up to 12 cycles.
  Interventions: Drug: Abiraterone acetate; Drug: Abiraterone acetate MTD; Drug: Dexamethasone

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone 250 mg (1 capsule) up to 2000 mg (8 capsules) once daily, each dose will be tested in sequential order for 28 days to determine the MTD.
  Other Names: CB7630
Drug: Abiraterone acetate MTD — Abiraterone acetate MTD orally for 12 cycles (28 day each).
  Other Names: CB7630
Drug: Dexamethasone — Dexamethasone 0.5 mg orally will be given (If participants have disease progression) daily up to 12 cycles.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and evaluate the safety, tolerability, and activity at the recommended dose (maximum tolerated dose [MTD]) of abiraterone acetate (also known as CB7630) in participants with hormone refractory prostate (gland that makes fluid that aids movement of sperm) cancer (HRPC).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) study to evaluate the safety, tolerability, and recommended dose of abiraterone acetate taken orally (by mouth), once daily in participants with HRPC. The study will consist of a dose escalation stage (Phase 1) that will be conducted to determine the MTD of abiraterone and an activity evaluation stage (Phase 2) to evaluate the activity of abiraterone in participants with HRPC. Escalated doses of abiraterone (starting at 250 milligram [mg] up to a maximum of 2000 mg) will be given for 28-day treatment periods to determine the MTD. Participants will be given MTD of abiraterone for up to 12 cycles (28 day each) in Phase 2 of the study. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically (pertaining to the disease status of body tissues or cells) documented adenocarcinoma of the prostate, clinically refractory (not responding to treatment) or resistant to hormone therapy, as documented by progression following at least one hormonal therapy
* Prostate specific antigen (PSA) evidence for progressive prostate cancer
* Participants who were withdrawn from anti-androgen therapy less than 6 months prior to inclusion in the study require one PSA higher than the last pre-withdrawal PSA or 2 increases in PSA documented after the post-withdrawal nadir(value) greater than or equal to 4 weeks from treatment withdrawal if treated with flutamide and greater than or equal to 6 weeks if treated with bicalutamide or nilutamide
* Eastern Cooperative Oncology Group (ECOG) performance status score equal to 0 or 1
* Life expectancy of greater than or equal to12 week

Exclusion Criteria:

* Participants with central nervous system (the brain and spinal cord) disease and/or brain metastases
* No currently active second malignancy (cancer or other progressively enlarging and spreading tumor) other than non-melanoma skin cancer
* Myocardial infarction within the 6 months prior to start of study
* No active or uncontrolled autoimmune disease (disorder in which a person's immune system attacks parts of his or her own body) that may require corticosteroid therapy during protocol treatment
* Major surgery or significant traumatic injury within 4 weeks of start of study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology Clinical Trial, Study Director — Cougar Biotechnology, Inc.
Locations (1):
- Sutton, United Kingdom

REFERENCES:
- See also: NATIONAL CANCER INSTITUTE — http://www.cancer.gov/
- See also: PROSTATE CANCER — http://www.nlm.nih.gov/medlineplus/prostatecancer.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 250 mg/Day: Abiraterone acetate 250 milligram (mg) capsule administered orally daily for 28-day treatment period to determine the maximum tolerated dose (MTD) in Phase 1 of the study. Participants received MTD (1000 mg) of abiraterone acetate for 12 cycles (28 day each) in Phase 2 of the study. Dexamethasone 0.5 mg administered orally (if participants have disease progression) daily up to 12 cycles.
- 500 mg/Day: Abiraterone acetate 500 mg capsules (2 x 250 mg capsules) administered orally daily for 28-day treatment period to determine the MTD in Phase 1 of the study. Participants received MTD of abiraterone acetate for 12 cycles (28 day each) in Phase 2 of the study. Dexamethasone 0.5 mg administered orally (if participants have disease progression) daily up to 12 cycles.
- 750 mg/Day: Abiraterone acetate 750 mg capsules (3 x 250 mg capsules) administered orally daily for 28-day treatment period to determine the MTD in Phase 1 of the study. Participants received MTD of abiraterone acetate for 12 cycles (28 day each) in Phase 2 of the study. Dexamethasone 0.5 mg administered orally (if participants have disease progression) daily up to 12 cycles.
- 1000 mg/Day: Abiraterone acetate 1000 mg capsules (4 x 250 mg capsules) administered orally daily for 28-day treatment period to determine the MTD in Phase 1 of the study. Participants received MTD of abiraterone acetate for 12 cycles (28 day each) in Phase 2 of the study. Dexamethasone 0.5 mg administered orally (if participants have disease progression) daily up to 12 cycles.
- 2000 mg/Day: Abiraterone acetate 2000 mg capsules (8 x 250 mg capsules) administered orally daily for 28-day treatment period to determine the MTD in Phase 1 of the study. Participants received MTD of abiraterone acetate for 12 cycles (28 day each) in Phase 2 of the study. Dexamethasone 0.5 mg administered orally (if participants have disease progression) daily up to 12 cycles.
Period: Period 1 (Phase 1)
Arm/Group | 250 mg/Day | 500 mg/Day | 750 mg/Day | 1000 mg/Day | 2000 mg/Day
Started | 3 | 3 | 3 | 42 | 3
Completed | 2 | 2 | 3 | 25 | 2
Not Completed | 1 | 1 | 0 | 17 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 5 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 1 | 1 | 0 | 10 | 1
Not completed — Other | 0 | 0 | 0 | 1 | 0
Period: Period 2 (Phase 2)
Arm/Group | 250 mg/Day | 500 mg/Day | 750 mg/Day | 1000 mg/Day | 2000 mg/Day
Started | 1 (1 participant did not continue to Phase 2 of the study.) | 2 | 2 (1 participant did not continue to Phase 2 of the study.) | 23 (2 participants did not continue to Phase 2 of the study.) | 2
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 2 | 23 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 1
Not completed — Disease Progression | 0 | 2 | 2 | 17 | 1
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- 250 mg/Day: Abiraterone acetate 250 mg capsule administered orally daily for 28-day treatment period to determine the MTD in Phase 1 of the study. Participants received MTD of abiraterone acetate for 12 cycles (28 day each) in Phase 2 of the study. Dexamethasone 0.5 mg administered orally (if participants have disease progression) daily up to 12 cycles.
- Total: Total of all reporting groups
Arm/Group | 250 mg/Day | 500 mg/Day | 750 mg/Day | 1000 mg/Day | 2000 mg/Day | Total
Number analyzed (Participants) | 3 | 3 | 3 | 42 | 3 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.07) | 68.7 (10.41) | 76 (8.19) | 70.4 (7.42) | 68 (12.17) | 69.9 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 42 | 3 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Prostate Specific Antigen (PSA) Response at Week 12
Description: The PSA response was measured according to PSA working group (PSAWG) criteria. All participants achieving a fall in PSA of greater than 50 percent from baseline, which has been confirmed by a second measurement at least 4 weeks after initial documentation, fulfill criteria for confirmed PSA response.
Time Frame: Baseline, Week 12
Population: All participants who were enrolled in the study and received 1000 milligram abiraterone acetate therapy with or without dexamethasone (including participants who received 1000 mg AA monotherapy). Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Number; unit: Participants
Groups:
- 1000 mg AA Monotherapy: Participants received 1000 milligram (mg) abiraterone acetate (AA) without dexamethasone.
- 1000 mg AA Therapy: Participants received 1000 mg abiraterone acetate with or without dexamethasone.
Arm/Group | 1000 mg AA Monotherapy | 1000 mg AA Therapy
Number analyzed (Participants) | 11 | 29
Participants | 10 | 25

2. Secondary Outcome: Number of Participants With Objective Tumor Response
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as greater than or equal to 30 percent decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study greater than or equal to 4 weeks after initial documentation of response.
Time Frame: Baseline up to end of study (1160 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 1000 mg AA Therapy
Number analyzed (Participants) | 38
Participants
  Complete response | 0
  Partial response | 8

3. Secondary Outcome: Duration of Prostate Specific Antigen (PSA) Response
Description: Duration of PSA response in participants on abiraterone acetate therapy was measured as the duration between PSA 50 percent decline date and PSA progression date as defined by the PSAWG criteria.
Time Frame: Baseline up to end of study (1160 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | 1000 mg AA Therapy
Number analyzed (Participants) | 27
Days | 141 [85 to 235]

4. Secondary Outcome: Duration of Objective Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Number of participants with objective response based on assessment of confirmed CR or confirmed PR according to RECIST. Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as greater than or equal to 30 percent decrease in sum of the LD of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study greater than or equal to 4 weeks after initial documentation of response.
Time Frame: Baseline up to end of study (1160 days)
Population: Duration of response was not analyzed as majority of participants with objective tumor response were lost to follow-up.
Arm/Group | 1000 mg AA Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Disease Progression
Description: Disease progression was defined as greater than 25 percent increase in sum of longest diameter of target lesions compared to baseline.
Time Frame: Baseline up to end of study (1160 days)
Population: Data was not analyzed because at the time to progression, participants also received dexamethasone treatment, making it impractical to accurately define disease progression.
Arm/Group | 1000 mg AA Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Description: Overall survival was the duration from enrollment to death. For participants who are alive, overall survival was censored at the last contact.
Time Frame: Baseline up to end of study (1160 days)
Population: Data was not analyzed due to high number of participants censored for survival.
Arm/Group | 1000 mg AA Therapy
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Serum Blood Levels of Testosterone
Description: Concentration of testosterone in blood was measured in nanogram per deciliter (ng/dL).
Time Frame: Baseline, Cycle 2 (within 3 days prior to Day 29)
Population: All participants who were enrolled in the study and received 1000 mg abiraterone acetate therapy with or without dexamethasone (including participants who received 1000 mg AA monotherapy). Here 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable at specified time point.
Measure: Median (Full Range); unit: ng/dL
Arm/Group | 1000 mg AA Therapy
Number analyzed (Participants) | 28
ng/dL
  Baseline (n = 23) | 3 [1 to 10]
  Cycle 2 (n = 28) | 1 [1 to 186]

8. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 30 days after the last dose of study medication
Population: Included all participants who received any amount of the study medication.
Measure: Number; unit: participants
Arm/Group | 250 mg/Day | 500 mg/Day | 750 mg/Day | 1000 mg/Day | 2000 mg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 42 | 3
participants
  AEs | 3 | 3 | 3 | 41 | 3
  SAEs | 2 | 2 | 0 | 20 | 2

9. Other Pre Specified Outcome: Serum Blood Levels of Testosterone Precursors
Description: Concentration of Cortisol, Aldosterone, Corticosterone, 11-Deoxycortisol, Deoxycorticosterone and Dehydroepiandrostenedione Sulphate (DHEA-S) in blood was measured in nanogram per deciliter (ng/dL).
Time Frame: Baseline, Cycle 2 (within 3 days prior to Day 29)
Population: as for outcome 7
Measure: Median (Full Range); unit: ng/dL
Arm/Group | 1000 mg AA Therapy
Number analyzed (Participants) | 33
ng/dL
  Cortisol; Baseline (n = 33) | 12000 [7000 to 23000]
  Cortisol; Cycle 2 (n = 29) | 4000 [1000 to 11000]
  Aldosterone; Baseline (n=33) | 8 [1 to 32]
  Aldosterone; Cycle 2 (n=29) | 8 [1 to 61]
  Corticosterone; Baseline (n=33) | 193 [4 to 1041]
  Corticosterone; Cycle 2 (n=27) | 6797 [12 to 17148]
  11-Deoxycortisol; Baseline (n=31) | 39 [20 to 233]
  11-Deoxycortisol; Cycle 2 (n=25) | 73 [20 to 836]
  Deoxycorticosterone; Baseline (n=32) | 6 [2 to 31]
  Deoxycorticosterone; Cycle 2 (n=28) | 121 [33 to 1627]
  DHEA-S; Baseline (n=32) | 30000 [15000 to 176000]
  DHEA-S; Cycle 2 (n=28) | 15000 [15000 to 15000]

10. Other Pre Specified Outcome: Time to Prostate Cancer Pain Progression
Description: The time from start of study treatment to the development/worsening of pain due to prostate cancer requiring one or more of the following treatments: 1- Opioid therapy (therapy with morphine like medicines for 10 out of 14 consecutive days); 2- Glucocorticoid therapy; 3- Initiation of >= 5 mg of prednisolone for 10 out of 14 consecutive days; 4- Radionuclide therapy; 5- Radiation therapy (x-ray or cobalt treatment); 6- Chemotherapy (treatment of disease by chemical agents). Participants who do not experience prostate cancer pain were censored on their last day on study. Time to prostate cancer pain progression was measured by Kaplan-Meier method.
Time Frame: Baseline up to 12 cycles
Population: Median time was not reached as data was not matured at the time of the analysis, hence no data could be reported.
Arm/Group | 1000 mg AA Therapy
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Number of Participants With Change From Baseline in Biochemical Bone Markers
Time Frame: Baseline, Cycle 2, 4, 8, 12
Population: Data was reported in individual participant listings but not summarized due to statistical constraints.
Arm/Group | 1000 mg AA Therapy
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Mean Plasma Concentration of Abiraterone
Time Frame: Pre-dose on Day 1, 8 and 15 of Cycle 1, Day 1 of Cycle 2, Day 1 of Cycle 3; 1, 2, 4, 6, 8, 24, 48 and 72 hours after first dose was given
Population: Data was not statistically summarized but reported in individual participant listing as per planned analysis.
Groups:
- Abiraterone Acetate 250 mg: Abiraterone acetate 250 mg capsule given orally daily for 28-day treatment period to determine the maximum tolerated dose (MTD) in Phase 1 of the study.
- Abiraterone Acetate 500 mg: Abiraterone acetate 500 mg capsules (2 x 250 mg capsules) given orally daily for 28-day treatment period to determine the maximum tolerated dose (MTD) in Phase 1 of the study.
- Abiraterone Acetate 750 mg: Abiraterone acetate 750 mg capsules (3 x 250 mg capsules) given orally daily for 28-day treatment period to determine the maximum tolerated dose (MTD) in Phase 1 of the study.
- Abiraterone Acetate 1000 mg: Abiraterone acetate 1000 mg capsules (4 x 250 mg capsules) orally daily given for 28-day treatment period to determine the maximum tolerated dose (MTD) in Phase 1 of the study.
- Abiraterone Acetate 2000 mg: Abiraterone acetate 2000 mg capsules (8 x 250 mg capsules) given orally daily for 28-day treatment period to determine the maximum tolerated dose (MTD) in Phase 1 of the study.
Arm/Group | Abiraterone Acetate 250 mg | Abiraterone Acetate 500 mg | Abiraterone Acetate 750 mg | Abiraterone Acetate 1000 mg | Abiraterone Acetate 2000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax) of Abiraterone
Description: The Cmax is defined as maximum observed analyte concentration.
Time Frame: as for outcome 12
Population: Included all participants who enrolled into the study regardless of the amount of the trial medication received. Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Abiraterone Acetate 250 mg | Abiraterone Acetate 500 mg | Abiraterone Acetate 750 mg | Abiraterone Acetate 1000 mg | Abiraterone Acetate 2000 mg
Number analyzed (Participants) | 3 | 3 | 2 | 9 | 3
nmol/L | 219 (172.77) | 284 (132.38) | 1032 (344.01) | 571 (443.18) | 531 (219.02)

14. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Abiraterone
Description: The Tmax is defined as actual sampling time to reach maximum observed plasma concentration. The analyte concentration associated with Tmax is referred to as Cmax.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Abiraterone Acetate 250 mg | Abiraterone Acetate 500 mg | Abiraterone Acetate 750 mg | Abiraterone Acetate 1000 mg | Abiraterone Acetate 2000 mg
Number analyzed (Participants) | 3 | 3 | 2 | 9 | 3
hours | 2.050 (0.02) | 2.588 (1.02) | 1.709 (0.41) | 3.159 (1.79) | 2.672 (1.14)

15. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Abiraterone
Description: Area under the plasma concentration time-curve from time zero to the last quantifiable concentration (AUClast).
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours*nmol/L
Arm/Group | Abiraterone Acetate 250 mg | Abiraterone Acetate 500 mg | Abiraterone Acetate 750 mg | Abiraterone Acetate 1000 mg | Abiraterone Acetate 2000 mg
Number analyzed (Participants) | 3 | 3 | 2 | 9 | 3
hours*nmol/L | 1253 (519.78) | 1334 (731.47) | 4294 (1295.20) | 4371 (3427.54) | 4754 (1659.13)

16. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Abiraterone
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours*nmol/L
Arm/Group | Abiraterone Acetate 250 mg | Abiraterone Acetate 500 mg | Abiraterone Acetate 750 mg | Abiraterone Acetate 1000 mg | Abiraterone Acetate 2000 mg
Number analyzed (Participants) | 3 | 3 | 2 | 9 | 3
hours*nmol/L | 1369 (505.39) | 1448 (749.01) | 4537 (1333.42) | 4615 (3660.48) | 4983 (1755.24)

17. Other Pre Specified Outcome: Plasma Decay Half-Life (t1/2) of Abiraterone
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Abiraterone Acetate 250 mg | Abiraterone Acetate 500 mg | Abiraterone Acetate 750 mg | Abiraterone Acetate 1000 mg | Abiraterone Acetate 2000 mg
Number analyzed (Participants) | 3 | 3 | 2 | 9 | 3
hour | 11.6 (10.14) | 9.5 (7.02) | 10.8 (5.91) | 10.6 (4.69) | 12.0 (2.29)

18. Other Pre Specified Outcome: Time to Last Quantifiable Plasma Concentration (Tlast) of Abiraterone
Description: The actual sampling time of last measurable (non-below the limit of quantification [BQL]) analyte concentration. The analyte concentration associated with Tlast is referred to as Clast.
Time Frame: as for outcome 12
Population: Data was not statistically summarized but reported in individual participant listing as per planned analysis.
Arm/Group | Abiraterone Acetate 250 mg | Abiraterone Acetate 500 mg | Abiraterone Acetate 750 mg | Abiraterone Acetate 1000 mg | Abiraterone Acetate 2000 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 250 mg/Day | 500 mg/Day | 750 mg/Day | 1000 mg/Day | 2000 mg/Day
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 0/3 | 20/42 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 41/42 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg/Day (N=3) | 500 mg/Day (N=3) | 750 mg/Day (N=3) | 1000 mg/Day (N=42) | 2000 mg/Day (N=3)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg/Day (N=3) | 500 mg/Day (N=3) | 750 mg/Day (N=3) | 1000 mg/Day (N=42) | 2000 mg/Day (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 11 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 9 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 2 | 5 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 8 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 1 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 21 | 2
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 4 | 0
Injection site discolouration (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 19 | 3
Pitting oedema (General disorders) | 0 | 0 | 0 | 2 | 2
Pyrexia (General disorders) | 1 | 1 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Gingival infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 5 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 3 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 8 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 5 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 3 | 0
Blood acid phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 0
Blood creatine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 3 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 6 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 34 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 12 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 8 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 5 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 9 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 7 | 2
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 6 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 5 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 5 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 4 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0
Pyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 3 | 0
Testicular atrophy (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 8 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1 | 6 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 15 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less